CLINICAL TRIAL: NCT04573556
Title: Multicenter, Post-marketing Observational (Non-interventional) Study to Evaluate the Safety of DAYVIGO Tablet in Patients With Insomnia.
Brief Title: A Study to Evaluate the Safety of DAYVIGO (Lemborexant) Tablets in Participants With Insomnia.
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2006-M081-501
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-09

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: E2006; Lemborexant; Insomnia; Non-interventional; Dayvigo
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lemborexant: Participants with insomnia will initiate treatment with lemborexant 5 milligram (mg), tablet, orally as per the clinical judgment of the treating physician as part of routine clinical care. Dosage and administration of lemborexant tablet will be according to package insert and actual dosing and frequency will be decided by physician including dose escalation from initial dose of 5 mg up to 10 mg once daily. All participants will be observed prospectively for up to 24 weeks.
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — Lemborexant oral tablets.
  Other Names: E2006; DAYVIGO

SUMMARY:
The purpose of the study is to evaluate the incidence of somnolence, parasomnia, narcoleptic symptoms, and suicidal ideation/suicidal behavior after administration of lemborexant (DAYVIGO) in daily practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are treated with lemborexant
2. Participants who provide consent for participation in the study
3. Participants who were registered in EDC by 14 days after DAYVIGO treatment initiation

Exclusion Criteria:

1. Participants who were enrolled in this study before obtaining informed consent of this study
2. Participants who were participating in a clinical trial at the time of this study

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 300 participants with insomnia
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | Up to 24 Weeks
  The adverse events considered by the investigators to be related to treatment with lemborexant will be classified as ADRs. The incidence of somnolence, parasomnia symptoms (nightmare, abnormal dreams, exploding head syndrome etc.), narcoleptic symptoms (sleep paralysis, hypnagogic hallucination, hypnopompic hallucination and cataplexy etc.), and suicidal ideation/suicidal behavior (intentional overdose, self-injurious ideation, suicidal ideation etc.) will be determined.

SECONDARY OUTCOMES:
Number of Participants With Response to Treatment | Up to 24 Weeks
  Response to treatment will be assessed by the impression of general improvement consisting of "Improvement", "No change", and "Worsening". One of these ratings will be selected based on physician's impression according to participants' complaints of insomnia symptoms and will be recorded in Electronic Data Capture (EDC).

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Eisai trial site 1, Nagoya
  - Eisai trial site 2, Osaka
  - Eisai trial site 3, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.